CLINICAL TRIAL: NCT00612118
Title: A Randomised, Double Blind, 2-way Crossover Trial of 8 Days Repeat Dosing With Intranasal GSK256066 and Azelastine Hydrochloride in the Vienna Challenge Chamber in Subjects With Seasonal Allergic Rhinitis (SAR)
Brief Title: A Phase II Study Evaluating Intranasal GSK256066 and Azelastine Hydrochloride in Subjects With Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IPR110982
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2011-02

CONDITIONS: Allergic Rhinitis; Rhinitis, Allergic, Seasonal
Keywords: Allergic rhinitis,; Vienna Challenge Chamber
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal | interventions — 6-((3-((dimethylamino)carbonyl)phenyl)sulfonyl)-8-methyl-4-((3-methyloxyphenyl)amino)-3-quinolinecarboxamide; azelastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK256066 — 200mcg bd
Drug: azelastine hydrochloride — 140mcg
  Other Names: GSK256066

SUMMARY:
This study is an 8 day, randomised, double blind, 2-way crossover trial of repeat doses of intranasal GSK256066 and azelastine hydrochloride in the Vienna Challenge Chamber in subjects with seasonal allergic rhinitis (SAR). Laboratory safety assessments, 12-lead electrocardiograph (ECG), vital signs and adverse event enquiries will be made throughout the study. Nasal examination, symptom scores, and allergen challenge assessments will also be performed at various time points throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* The subject is healthy. Healthy subjects are defined as individuals who are free from clinically significant illness or disease as determined by their medical history (including family), physical examination, laboratory studies, and other tests.
* Male or female between 18 and 50 years inclusive.
* A female subject is eligible to participate if she is of:

  * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory].
  * Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the end of the study.
* Body mass index less than 29.0 kg/m² with weight range of 55.0kg (females 50kg) to 95.0kg inclusive.
* The subject has a history of seasonal allergic rhinitis.
* The subject exhibits a moderate response to 1500 grass pollen grains/m3 after 2 hours in the Vienna Challenge Chamber, defined as a nasal symptom score of at least 6. (Nasal symptom score is the sum of obstruction, rhinorrhoea, itch and sneeze, each of which have been scored on a scale from 0 to 3).
* The subject has a positive skin prick test (wheal ³ 4mm) for grass pollen at or within the 12 months preceding the screening visit.
* The subject has a positive RAST (³ class 2) for grass pollen at or within the 12 months preceding the screening visit.
* The subject is a current non-smoker who has not used any tobacco products in the 6 months preceding the screening visit with a pack history of £ 10 pack years.
* The subject must have a baseline FEV1>80% predicted and a baseline FEV1(maximum recorded value)/FVC(maximum recorded value)>70% predicted (using the Standardized Lung Function Testing guidelines produced by European Community for Coal and Steel)
* There are no conditions or factors which would make the subject unlikely to be able to stay in the chamber for 4 hours.
* The subject is capable of giving informed consent which includes compliance with the requirements and restrictions listed in the consent form
* The subject is available to complete all study measurements.

Exclusion Criteria:

* Pregnant or nursing females
* Women of childbearing potential who are unwilling or unable to use an appropriate method of contraception, as listed in Section 8.1, from at least two weeks prior to the first dose of study medication; and to continue until the end of the study.
* On examination the subject is found to have any structural nasal abnormalities or nasal polyposis, a history of frequent nosebleeds, recent nasal surgery or recent (within 3 weeks) or ongoing upper respiratory tract infection which in the Responsible Physician's opinion renders the subject unsuitable for participation in the study
* Any respiratory disease other than mild stable asthma that is controlled with occasional use of as-needed short-acting beta-agonists and associated with normal lung function.
* The subject is likely to be unable to abstain from salbutamol use for 8 hours before a challenge
* The subject has a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* The subject is concurrently participating in another clinical study or has participated in a study with an investigational product (new chemical entity) during the previous 4 months or in any clinical study during the previous month.
* The subject has a screening QTc(B) value >450msec, PQ interval outside the range 120 to 240msec or an ECG that is not suitable for QT measurements (e.g. poorly defined termination of the T-wave). In addition subjects will be excluded if they have a history of atrial and ventricular arrhythmia.
* A supine blood pressure that is persistently higher than 140/90 millimetres of mercury (mmHg) at screening.
* A supine mean heart rate outside the range 40-90 beats per minute (bpm) at screening.
* The subject has donated a unit of blood (450mL) within the previous 3 months or intends to donate within 3 months of completing the study.
* The subject is currently taking regular (or a course of) medication whether prescribed or not, including steroids, vitamins, macrolides, anti-fungal agents and herbal remedies (e.g. St. John's Wort). Paracetamol (£2g/day) and occasional as needed use of short-acting beta agonists is permitted.
* The subject has used prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potent enzyme inducer) or 5 half-lives (which ever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and Sponsor the medication will not interfere with the study procedures or compromise subject safety.
* The subject has used oral, injectable or dermal steroids within 5 weeks or intranasal and/or inhaled steroids within 1 week of the screening visit.
* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease*, haematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, bronchiectasis or pulmonary fibrosis).

  *subjects will require normal serum creatinine clearance values at screening [calculated from serum creatinine by a predicting equation using Cockcroft-Gualt formula]. If the creatinine clearance value is greater than the upper limit of normal as determined by the local laboratory reference range, the Investigator will determine whether this is a clinically significant finding that would preclude participation.
* The subject regularly drinks more than 28 units of alcohol in a week if male, or 21 units per week if female. One unit of alcohol is defined as a medium (125 ml) glass of wine, half a pint (250 ml) of beer or one measure (24 ml) of spirits.
* The subject is at risk of non-compliance with the study procedures/restrictions.
* The subject is infected with the Hepatitis B, Hepatitis C, or HIV virus.
* The subject has an elevated Troponin T above the normal range.
* The subject, as deemed by the Investigator has a clinically significant CK-MB value above the normal range.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Investigate effect of repeat intranasal doses of azelastine hydrochloride alone vs. GSK256066 + azelastine hydrochloride on nasal symptoms of allergic rhinitis provoked by spending 4h in the Vienna Challenge Chamber after morning dosing on Day 8. | spending 4h in the Vienna Challenge Chamber after morning dosing on Day 8.

SECONDARY OUTCOMES:
Weighted mean eye symptom score (watery eyes, itchy eyes, red eyes) | over 1-4 hours on Day 8.
Weighted mean global symptom score (sneeze, itch, rhinorrhoea, obstruction, cough, itchy throat, itchy ears, watery eyes, itchy eyes and red eyes) | over 1-4 hours on Day 8.
Weighted mean nasal airflow (measured using active anterior rhinomanometry) and secretion weight (measured by weighing tissues) | over 1-4 hours on Day 8.
Weighted mean components of TNSS (sneeze, itch, rhinorrhoea and obstruction) | over 1-4 hours on Day 8.
FEV1, ECGs, Vital signs, AEs, and laboratory safety parameters.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Vienna, Austria